CLINICAL TRIAL: NCT01197040
Title: Low Steroid Dose Combined With Mycophenolic Acid (Myfortic) Compared With High Dose Steroid for Minimal Change Nephrotic Syndrome
Brief Title: Evaluation of Low Dose Corticosteroids Efficiency, Associated With Myfortic ® in the Treatment of Nephrotic Syndrome
Acronym: MSN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P071226
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2015-10

CONDITIONS: Nephrotic Syndrome
Keywords: Minimal Change Nephrotic Syndrome; Complete remission; Myfortic; Minimal Change Disease
MeSH Terms: conditions — Nephrotic Syndrome; Nephrosis, Lipoid; Pathologic Complete Response | interventions — Prednisone; Mycophenolic Acid; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B-Experimental (Experimental): Experimental
  Interventions: Drug: acid mycophenolic (Myfortic)
- A-Active Comparator (Active Comparator): Active Comparator
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — 1 mg/kg/day for 4 weeks. Then, the dose will be progressively tapered if the remission will be achieved. For patients who exhibit incomplete remission at this time, high dose steroid will be continued for 4 weeks again before the tapering.
  Other Names: Monotherapy: treatment with only corticosteroids at doses usually 1 mg/kg/day,following a plan of reduction based on the degree of remission.
  Arms: A-Active Comparator
Drug: acid mycophenolic (Myfortic) — patients will receive prednisone 0.5 mg/kg/day combined with mycophenolic acid (MyforticR) 1440 mg/day. The management of steroid therapy will be identical in both groups, while MyforticR will be continued for six months
  Other Names: Bitherapy: Association of low dose corticosteroids 0.5 mg/kg/day and Myfortic ® at a dose of 1440 mg/day.
  Arms: B-Experimental

SUMMARY:
A multicenter, randomized, study will be performed to evaluate the efficacy of low dose steroid combined with mycophenolic acid (MyforticR) versus high dose steroid in inducing remission in adults with minimal change nephrotic syndrome (MCNS). One hundred and fourteen patients (CPP decision 2009-04-02-a5) will be included in this study. They will be randomly assigned to an open label treatment with either prednisone

1 mg/kg/day (arm A) or 0,5 mg/kg/day plus myforticR 1440 mg/day (arm B) for four weeks. The outcome will be compared during one-year follow up

DETAILED DESCRIPTION:
The treatment for minimal change nephrotic syndrome (MCNS) is empirically based on high dose steroid. However, the side effects in adult patients are often significant and induce a lot of complications. This prospective study aimed to compare low dose steroid combined with mycophenolic acid (MyforticR) versus high dose steroid in the treatment of the first episode of MCNS.

Treatment Plan

After baseline evaluation including clinical biological and histological analyses, all eligible patients will be an open label assigned to two groups:

Group A: patients will receive prednisone 1 mg/kg/day for 4 weeks. Then, the dose will be progressively tapered if the remission will be achieved. For patients who exhibit incomplete remission at this time, high dose steroid will be continued for 4 weeks again before the tapering.

Group B: patients will receive prednisone 0.5 mg/kg/day combined with mycophenolic acid (MyforticR) 1440 mg/day. The management of steroid therapy will be identical in both groups, while MyforticR will be continued for six months.

In both groups, patients who will not achieve remission after 8 weeks of steroid therapy at full dose will be excluded from the study.

Statistical Analysis In this multicenter, randomized trial, the primary and secondary end points will be the rate of complete remission within 4 and 8 weeks of the start of induction therapy, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic nephrotic syndrome
* Flare of idiopathic syndrome without treatment from one year
* Confirming by Renal Biopsy

Exclusion Criteria:

* Secondary nephrotic syndrome
* Pregnancy
* Focal Segmental Glomerular sclerosis lesion in the Biopsy
* Neutropenia < 2000/mm3
* Hb<9gr/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2009-10; Primary Completion 2014-07 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
complete remission | within 4 weeks
  complete remission

SECONDARY OUTCOMES:
complete remission | within 8 weeks
  complete remission
partial remission | within 4 and 8 weeks
  partial remission
Adverse effects in both arms | 1 year
  Adverse effects in both arms
Number of flare in both arms | at 1 year
  Number of flare in both arms

CONTACTS AND LOCATIONS:
Overall Officials: Philippe REMY, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, Val de Marne, France

REFERENCES:
- [Derived] Azukaitis K, Palmer SC, Strippoli GF, Hodson EM. Interventions for minimal change disease in adults with nephrotic syndrome. Cochrane Database Syst Rev. 2022 Mar 1;3(3):CD001537. doi: 10.1002/14651858.CD001537.pub5. PMID 35230699
- [Derived] Remy P, Audard V, Natella PA, Pelle G, Dussol B, Leray-Moragues H, Vigneau C, Bouachi K, Dantal J, Vrigneaud L, Karras A, Pourcine F, Gatault P, Grimbert P, Ait Sahlia N, Moktefi A, Daugas E, Rigothier C, Bastuji-Garin S, Sahali D; MSN Trial Investigators. An open-label randomized controlled trial of low-dose corticosteroid plus enteric-coated mycophenolate sodium versus standard corticosteroid treatment for minimal change nephrotic syndrome in adults (MSN Study). Kidney Int. 2018 Dec;94(6):1217-1226. doi: 10.1016/j.kint.2018.07.021. Epub 2018 Oct 29. PMID 30385039